CLINICAL TRIAL: NCT04746833
Title: Development and Pilot Testing of LIMIT: a Multicomponent Tool to Support Opioid Tapering
Brief Title: Development/Testing of SUMMIT: a Tool to Help Patients Manage Pain While Tapering Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 17-228
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain
Keywords: m-health
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: We will conduct a 9-month, randomized, two-arm, parallel, open-label, feasibility trial. Eligible participants will be randomized to LIMIT versus a pain monitoring app. Outcome measures will be collected over 9 months.
  To ensure rigor and successful future implementation, we will: 1) develop an evidence based program with features proven to maximize engagement and retention; 2) ensure that the program includes mechanisms to address the diverse obstacles veterans report when consider opioid tapering (e.g. fear of pain flares and abandonment by the system); 3) employ a User Centered Design - with meaningful input from veterans and primary care providers throughout the development and testing phases; and 4) adhere to recently published guidelines for mobile health interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUMMIT (Experimental): Participants randomized to the experimental intervention will participate in a Motivational Interviewing (MI) session lasting between 30 and 60 minutes with study psychologist. All MI sessions will be audiotaped using a VA-approved digital recorder and transcribed verbatim. Participants will subsequently be shown how to access SUMMIT via a set of unique anonymized login credentials and to navigate the components of SUMMIT on one or more devices, depending on their preference. They will then be trained on how to complete the outcome surveys.
  Interventions: Behavioral: SUMMIT
- control (Placebo Comparator): Participants randomized to the control intervention will use an eHealth comparator: My Pain Diary: Chronic Pain Management (iPhone, Android). This app includes a pain monitoring functioning only, and thus will only minimally overlap, if at all, with SUMMIT's components. Control participants will not participate in a MI session. Participants will download the app and be shown how to use the My Pain Diary app and trained how to complete the outcome surveys
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: SUMMIT — multicomponent web-based application focused on pain self-management skills
  Arms: SUMMIT
Behavioral: control — My Pain Diary app
  Arms: control

SUMMARY:
There are nearly one million veterans being treated with long-term opioid therapy (LTOT) for chronic pain. Numerous short and long-term harms associated with LTOT and mounting evidence suggest they have modest or no benefit. Yet, currently available resources to support veterans to taper are inadequate. Primary care, where most LTOT in VHA is prescribed, is overburdened and straining to meet the challenge of caring for patients with chronic pain. A scalable, relatively inexpensive tapering intervention to support primary care and/or to extend the reach of resource-intensive specialty clinics would be of great benefit to veterans who are not deriving sufficient benefit from LTOT. As such, the goal of this study is to develop and test an interactive, theory-informed, multi-component mobile website to enable veterans to safely taper opioids while managing their pain.

DETAILED DESCRIPTION:
The investigators will conduct a 9-month, randomized, two-arm, parallel, open-label, feasibility trial of the multicomponent mobile website called SUMMIT. Eligible participants will be randomized to SUMMIT versus a pain monitoring app. Outcome measures will be collected over 9 months.

To ensure rigor and successful future implementation, the investigators will: 1) develop an evidence based program with features proven to maximize engagement and retention; 2) ensure that the program includes mechanisms to address the diverse obstacles veterans report when consider opioid tapering (e.g. fear of pain flares and abandonment by the system); 3) employ a User Centered Design - with meaningful input from veterans and primary care providers throughout the development and testing phases; and 4) adhere to recently published guidelines for mobile health interventions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Veterans will be primary care patients who are dispensed 84 consecutive days of a stable dose of opioids (reflecting three consecutive 28-day prescriptions) through primary care and who report stable levels of pain intensity over the past month.

Exclusion Criteria:

Exclusion criteria will be Veterans on liquid methadone or buprenorphine for opioid use disorder (OUD) and those who have transitioned to buprenorphine (transdermal or sublingual) for chronic pain, have hearing or visual impairments (not corrected with hearing aids or glasses), psychiatric conditions, cognitive impairments, or participating in a concurrent pain or opioid-related research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Becker, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (4):
- United States (4):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Becker WC. "Clues" That Patients May Be Willing to Consider Opioid Reductions. J Gen Intern Med. 2020 Jun;35(6):1629-1630. doi: 10.1007/s11606-020-05712-6. No abstract available. PMID 32221855

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SUMMIT | Control
Started | 24 | 20
Completed | 24 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUMMIT | Control | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.9) | 68.8 (9.3) | 65.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 21 | 16 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 8 | 4 | 12
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 20 | 44
Prescribed Opioids Difficulties Scale - Opioid Control Concerns [Mean (Standard Deviation); unit: units on a scale] — The PODS Control Concerns sub-scale includes 7 difficulties attributed to opioid use. Items range from 0 to 4 for a scale range from 0 to 28. Higher scores indicate that patients attributed more problems to their use of opioid medications.
  units on a scale | 6.3 (3.4) | 7.5 (4.1) | 6.9 (3.7)
Prescribed Opioids Difficulties Scale - Psychosocial Problems [Mean (Standard Deviation); unit: units on a scale] — The PODS Psychosocial Problems sub-scale includes 7 difficulties attributed to opioid use. Items range from 0 to 4 for a scale range from 0 to 28. Higher scores indicate that patients attributed more problems to their use of opioid medications.
  units on a scale | 7.5 (6.7) | 7.1 (6.0) | 7.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Daily Morphine Milligram Equivalents (MME)
Description: Morphine milligram equivalents per day based on participant self report.
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents per day
Arm/Group | SUMMIT | Control
Number analyzed (Participants) | 20 | 19
Morphine milligram equivalents per day | 25.1 (44.7) | 21.9 (28.6)
Statistical Analysis 1: Comparison: SUMMIT vs Control; Test type: Equivalence — mean of Summit will be equal to mean of control; p = .91, t-test, 2 sided

2. Primary Outcome: Minutes of Summit App Use
Description: Total number of minutes of use of the Summit app over the 6 month intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Minutes of use
Arm/Group | SUMMIT
Number analyzed (Participants) | 24
Minutes of use | 20.9 (19.8)
Statistical Analysis 1: Comparison: SUMMIT; descriptive statistic of system use; Test type: Other; simple descriptive findings for evaluation of feasibility of the Sumit app

3. Secondary Outcome: Behavior Intervention Rating Scale (BIRS)
Description: The BIRS is a 24-item validated measure of an intervention's acceptability and perceived effectiveness scored on 5-point agreement scales. The total score is divided by the total number of completed items and this ranges from 1 to 5. Higher mean item scores represent higher acceptability.
Time Frame: six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUMMIT | Control
Number analyzed (Participants) | 19 | 17
score on a scale | 4.4 (0.4) | 4.5 (0.4)
Statistical Analysis 1: Comparison: SUMMIT vs Control; Test type: Equivalence — standard null hypothesis of no difference between groups; p = .50, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 9 months
Description: Adverse events were defined as events related to the study.
Arm/Group | SUMMIT | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 0/24 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT04746833/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT04746833/ICF_000.pdf